CLINICAL TRIAL: NCT01383564
Title: Effect of Nasal Continuous Positive Airway Pressure in Uncontrolled Nocturnal Asthmatic Patients With Moderate Obstructive Sleep Apnea Syndrome
Brief Title: Continuous Positive Airway Pressure Use in Asthma With Moderate to Severe Obstructive Sleep Apnea Patients
Acronym: OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Honorary Clinical Tutor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asthma OSA/Ng/2011
Record Dates: First submitted 2011-06-10; First posted 2011-06-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: OSA

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP group (Active Comparator): CPAP group
  Interventions: Procedure: CPAP group
- non CPAP group (Placebo Comparator): non CPAP group
  Interventions: Procedure: non CPAP group

INTERVENTIONS:
Procedure: CPAP group — Patients will be given a CPAP education program by our respiratory nurse supplemented by education brochure and a video. Attended overnight CPAP titration will be performed with the auto-titrating device. The CPAP level for each patient in the therapeutic CPAP arm is set at the minimum pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night as determined by the overnight CPAP titration study. Patients in the CPAP therapy will be provided careful mask-fitting, chin strap to prevent mouth leak, regular review by our nurses, a basic CPAP device with intrinsic time clock to monitor CPAP usage and standard stroke rehabilitation programme. Patients on conservative treatment will only be offered standard treatment for asthma
  Other Names: CPAP intervention group
  Arms: CPAP group
Procedure: non CPAP group — Patients who are randomised to non CPAP group will receive general health advice and no CPAP therapy will be arranged for them during the study period.
  Other Names: No CPAP given
  Arms: non CPAP group

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) and asthma are both common disorders in Hong Kong, with prevalence of at least 4% among the middle-aged male Hong Kong (HK) Chinese populations and 7.2% in young adults respectively. OSAS is characterized by repetitive episodes of upper airway obstruction, causing intermittent hypoxia, sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor health status. Continuous positive airway pressure (CPAP) is the first line of therapy for sleep apnea. CPAP provides a pneumatic stent for the upper airway, eliminating the airway collapse during inspiration.

Asthma is a chronic inflammatory disorder of airways, characterized by airway hyperresponsiveness that leads to recurrent episodes of wheezing, breathless, chest tightness, and coughing, particularly at night or in the early morning. Nocturnal asthma is not a different condition from asthma and is defined as a variable worsening of asthma at night, in which the mechanisms are not completely understood.

The prevalence of OSAS in asthmatic patients has not yet been studied, but several studies have reported an increased prevalence of OSAS symptoms in asthmatic patients. OSAS and asthma share some common risk factors, which include obesity, gastroesophageal reflux and rhinitis. CPAP treatment has been shown in prospective clinical studies to have a positive impact on asthma outcome in patients with concomitant OSAS, for example, improvement of asthma related quality of life in subjects with stable mild-to-moderate asthma, but there was no change in the airway responsiveness or forced expiratory volume in one second. Although important, these studies included small numbers of participants used nonrandomized designs. This study is to assess the impact of CPAP treatment on asthma control among patients with nocturnal symptoms and moderate OSAS.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) and asthma are both common disorders in Hong Kong, with prevalence of at least 4% among the middle-aged male Hong Kong (HK) Chinese populations and 7.2% in young adults respectively. OSAS is characterized by repetitive episodes of upper airway obstruction, causing intermittent hypoxia, sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor health status. Continuous positive airway pressure (CPAP) is the first line of therapy for sleep apnea. CPAP provides a pneumatic stent for the upper airway, eliminating the airway collapse during inspiration.

Asthma is a chronic inflammatory disorder of airways, characterized by airway hyperresponsiveness that leads to recurrent episodes of wheezing, breathless, chest tightness, and coughing, particularly at night or in the early morning. Nocturnal asthma is not a different condition from asthma and is defined as a variable worsening of asthma at night, in which the mechanisms are not completely understood. It may be driven by circadian rhythms of circulating hormones such as epinephrine, cortisol, and melatonin and neural mechanisms such as cholinergic tone. An increase in airway inflammation at night has been reported. This might reflect a reduction in endogenous anti-inflammatory mechanisms. Other factors that have been proposed as possible causes for overnight bronchoconstriction are interruption of bronchodilator or other treatment, allergens in bedding, airway cooling, supine posture, and gastroesophageal reflux (GER).

Prevalence of OSAS in asthma: The prevalence of OSAS in asthmatic patients has not yet been studied, but several studies have reported an increased prevalence of OSAS symptoms in asthmatic patients. Large epidemiologic studies demonstrated that asthma patients are more frequently report snoring. In a longitudinal study, asthma was an independent risk factor for development of snoring. OSAS symptoms are highly prevalent in clinic-based populations of well-characterized asthma patients. Polysomnography revealed high frequencies of OSAS (88% and 95.5%) in patients with difficult-to-control asthma.

Common risk factors contributing OSAS asthma: OSAS and asthma share some common risk factors. Fifty percent of the obese in Caucasian populations have OSAS, and among those with OSAS, 40% are obese. However, in a community study of sleep-disordered breathing in middle-aged Chinese men in Hong Kong, the average body mass index (BMI) of habitual snorer was 25.1 kg/m2 and that of OSAS was 27kg/m2, making the contribution of obesity in OSAS less as important as in the western counterpart. Apart from obesity, the prevalence of GER is increased in patients with OSAS. It has been suggested that obesity contributes to the same risk factors for OSAS and GER. However, OSAS patients exhibit significantly more GER than do members of the average population even when one controls for alcohol intake and BMI. GER occurring during sleep is a well-known trigger for nocturnal asthma and can provoke asthma symptoms through vagal reflexes induced by exposure of the esophagus to acid. OSAS-induced acid reflux may play a causative role in triggering asthma symptoms. Another possible etiology for the high prevalence of OSAS symptoms in asthmatic patients is the increased incidence of nasal obstruction in asthmatic patients. The nose is preferred breathing route during sleep, and nasal obstruction contributes to sleep disordered breathing in predisposed individuals. Rhinitis and chronic sinusitis are common conditions that may cause nasal congestion and consequently contribute to upper airway obstruction in OSAS.

The effect of CPAP treatment on asthma control:

CPAP treatment has been shown in prospective clinical studies to have a positive impact on asthma outcome in patients with concomitant OSAS. Although important, these studies included small numbers of participants used nonrandomized designs.

We hypothesize that OSAS contribute to the symptoms related to nocturnal asthma and that CPAP therapy would improve the asthma symptoms, airway hyperactivity and quality of life in patients with nocturnal asthma and OSAS. We aim to assess (1) asthma control, airway responsiveness, daytime sleepiness, cognitive function and health status at baseline and at 3 months after nasal CPAP treatment among our asthma patients with nocturnal symptoms and OSAS; (2) the acceptance and compliance of nasal CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* at least one nocturnal awakening or early morning awakening caused by asthmatic symptoms (cough, wheeze, chest tightness, and breathlessness)
* habitual snoring; able to give consent for joining the study

Exclusion Criteria:

* active smoking or quit smoking <6 months or smoking history >10 pack-years
* Cardiac failure
* cerebrovascular disease
* lung disease except asthma
* dementia or poor hand function that would inhibit the patients cooperating the sleep study or CPAP treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Asthma control test score | 3 months
  All patients with moderate OSAS will be assessed by an easy assessment tool for asthma control, known as the Asthma Control Test (ACT). It is a validated questionnaire in which various studies have proved its correlation with the clinical asthma control. The ACT consisted of five items; for each item, five options are provided pertaining to asthma control during the past 4 weeks. Each item is scored according to a 5-point scale, and the item scores are totalled for assessing asthma control, with higher total scores indicating better asthma control.

SECONDARY OUTCOMES:
Spirometry | 3 months
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The most important aspects of spirometry are the forced vital capacity (FVC), which is the volume delivered during an expiration made as forcefully and completely as possible starting from full inspiration, and the forced expiratory volume in one second(FEV1), which is the volume delivered in the first second of an FVC manoeuvre. The value of FEV1 and FVC will be monitored in baseline and 3 months.
Epworth Sleepiness Score (ESS) | 3 months
  The Epworth Sleepiness Scale (ESS) is a questionnaire for assessing daytime sleepiness. It was first described in 1991 as a simple, self-administered questionnaire. The questionnaire is based on eight common situations in life. Subjects are asked to rate on a scale of 0-3 about how likely they would fall asleep or doze off in these circumstances. This gives a total score of 0 to 24 in each subject.
SF 36 questionnaire | 3 months
  The Short Form Health Survey (SF-36) is a survey of patient health. It is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.
Bronchial challenge test | 3 months
  A bronchial challenge test is one method of assessing airway responsiveness in which patient breathes in nebulised methacholine and then will be assessed by measuring the Forced Expiratory Volume in one second (FEV1).

CONTACTS AND LOCATIONS:
Overall Officials: Susanna SS Ng, MBChB, Principal Investigator — Chinese Univesrity of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng SSS, Chan TO, To KW, Chan KKP, Ngai J, Yip WH, Lo RLP, Ko FWS, Hui DSC. Continuous positive airway pressure for obstructive sleep apnoea does not improve asthma control. Respirology. 2018 Nov;23(11):1055-1062. doi: 10.1111/resp.13363. Epub 2018 Jul 10. PMID 29992713